CLINICAL TRIAL: NCT00757172
Title: A Phase II Study of Neoadjuvant Therapy With Cisplatin, Docetaxel, Panitumumab Plus Radiation Therapy Followed by Surgery in Patients With Locally Advanced Adenocarcinoma of the Distal Esophagus
Brief Title: Panitumumab, Docetaxel, Cisplatin, Radiation Therapy, and Surgery in Treating Patients With Newly Diagnosed, Locally Advanced Esophageal Cancer or Cancer of the Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z4051; ACOSOG-Z4051; CDR0000596674 (Registry Identifier: Physician Data Query); NCI-2009-00346 (Registry Identifier: NCI Clinical Trials Reporting Office); U10CA076001 (NIH)
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; adenocarcinoma of the gastroesophageal junction; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Panitumumab; Cisplatin; Docetaxel; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel + Cisplatin + Panitumumab + RT (Other): Patients received docetaxel (40 mg/m^2), cisplatin (40 mg/m^2) and panitumumab (6 mg/kg) on weeks 1, 3, 5, 7, and 9 with radiotherapy (RT) (5040 cGy, 180 cGy/day x 28 days) beginning week 5. Resection was planned after completing chemotherapy (CRT).
  Interventions: Biological: panitumumab; Drug: cisplatin; Drug: docetaxel; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: panitumumab
Drug: cisplatin
Drug: docetaxel
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to kill tumor cells or stop them from growing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with panitumumab and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving panitumumab together with docetaxel, cisplatin, radiation therapy, and surgery works in treating patients with newly diagnosed, locally advanced esophageal cancer or cancer of the gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the pathologic complete response rate in patients with newly diagnosed, locally advanced adenocarcinoma of the distal esophagus or gastroesophageal junction treated with neoadjuvant panitumumab and combination chemoradiotherapy followed by surgery.

Secondary

* To determine the near-complete pathologic response rate in the primary tumor (≤ 10% residual viable cancer).
* To determine the overall survival and disease-free survival rates of these patients.
* To determine the safety profile of this regimen.

OUTLINE: Patients receive panitumumab IV over 1 hour, docetaxel IV over 1 hour, and cisplatin IV over 1-2 hours on day 1 in weeks 1, 3, 5, 7, and 9. Patients also undergo radiotherapy once daily 5 days a week beginning in week 5 and continuing for 5.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Beginning 6-9 weeks after completion of chemoradiotherapy, patients with no evidence of metastatic disease undergo esophagectomy.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year OR every 6 months for 3 years.

ELIGIBILITY:
1. ≥ 18 years old
2. ECOG/Zubrod Performance Status 0-1
3. Biopsy-proven resectable primary (nonrecurrent) adenocarcinoma of the distal esophagus or GE junction (Siewert Type I or II)

   * Siewert Type I: adenocarcinoma of the distal esophagus
   * Siewert Type II: adenocarcinoma of the esophago-gastric junction/real cardia
4. Pre-registration EUS, CT of chest and upper abdomen, and PET must support a clinical stage of T3N0M0, T2-3N1M0 or T2-3N0-1M1a (celiac adenopathy must be ≤ 2 cm by EUS). Clinically staged T1 tumors and T2N0M0 tumors are not eligible. N1 does not require biopsy/FNA. Note: Patients requiring a stent for nutrition must have staging examinations and scans completed before stent placement.
5. No definitive radiological evidence of distant metastases.
6. No pre-existing grade 2 or greater peripheral neuropathy (CTCAE v3) of any etiology.
7. Adequate bone marrow, hepatic and renal function prior to registration:

   * WBC ≥ 3,000/mm³
   * ANC ≥ 1,500/mm³
   * Platelet count ≥ 100,000/mm³
   * Hemoglobin ≥ 9.5 g/dL
   * Creatinine ≤ 1.5 mg/dL
   * Total bilirubin ≤ 3 mg/dL
   * AST (SGOT) ≤ 2.0 times upper limit of normal (ULN)
   * ALT (SGPT) ≤ 2.0 times ULN
   * Alkaline phosphatase ≤ 2.0 times ULN
   * Albumin ≥ 2.0 g/dL OR prealbumin ≥ 15 mg/dL
   * Magnesium ≥ lower limit of normal (LLN)
8. Patient must be evaluated before registration by medical oncologist, radiation oncologist and surgeon and deemed fit for protocol therapy and surgery.
9. No prior invasive malignancy, unless disease-free for ≥ 5 years prior to registration (Exceptions: non-melanoma skin cancer, in-situ cancers).
10. Non-pregnant and non-breast feeding. Female participants of child-bearing potential must have a negative urine or serum pregnancy test prior to registration. Perimenopausal participants must be amenorrheic ≥ 12 months to be considered not of childbearing potential. All patients of reproductive potential must agree to use an an effective method of birth-control while receiving study therapy and for six months after completion of therapy.
11. No prior chest or upper abdomen radiotherapy; prior therapy with cisplatin, docetaxel, panitumumab or other anti-EGFR therapy or prior esophageal or gastric surgery (Exception: prior surgery to treat reflux disease)
12. No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psyschiatric illness/social situations that would limit compliance with study requirements.
13. No history of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan
14. No history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Craig Lockhart, MD, Study Chair — Washington University School of Medicine
Locations (21):
- United States (21):
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Dayton, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Result] Lockhart AC, Reed CE, Decker PA, Meyers BF, Ferguson MK, Oeltjen AR, Putnam JB, Cassivi SD, Montero AJ, Schefter TE; American College of Surgeons Oncology Group. Phase II study of neoadjuvant therapy with docetaxel, cisplatin, panitumumab, and radiation therapy followed by surgery in patients with locally advanced adenocarcinoma of the distal esophagus (ACOSOG Z4051). Ann Oncol. 2014 May;25(5):1039-44. doi: 10.1093/annonc/mdu091. Epub 2014 Feb 20. PMID 24562448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy participants were recruited between January 2009 to July 2011 from 24 institutions.
Pre-assignment Details: Five participants were declared ineligible. One participant had a celiac lymph node >2 cm and one participant had two primary tumors. Liver lesions were noted and not investigated in one participant. Two participants had Siewert type III tumors. These five participants were excluded from all analysis except adverse events.
Period: Overall Study
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Started | 65
Completed | 54 (Participants underwent surgery.)
Not Completed | 11
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 3
Not completed — Progression | 4

BASELINE CHARACTERISTICS:
Population: All registered participants who have met the eligibility criteria.
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 65
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants]
  0= Asymptomatic and fully active | 37
  1= Symptomatic; fully ambulatory | 28
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 27.8 [17.7 to 53.5]
Tumor location (Siewert Type) [Number; unit: participants] — Siewert Type I= Adenocarcinoma of the distal esophagus; Siewert Type II= Adenocarcinoma of the esophagogastric junction/real cardia
  participants
    I | 36
    II | 29
Clinical T Stage [Number; unit: participants]
  T2 = Tumor invades muscularis propria | 7
  T3= Tumor invades adventitia | 58
Clinical N Stage [Number; unit: participants]
  N0= No regional lymph node metastasis | 13
  N1= Regional lymph node metastasis | 52
Clinical M Stage [Number; unit: participants]
  M0= No distant metastasis | 56
  M1a= Metastasis in celiac or cervical lymph nodes | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response Following Surgery
Description: Pathologic complete response (pCR) was defined as no viable residual tumor cells. A cellular residual mucin pools should be noted but also considered a pathologic complete response.
Time Frame: Post surgery
Population: All participants who have met the eligibility criteria that have signed a consent form and began treatment.
Measure: Number; unit: participants
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Number analyzed (Participants) | 54
participants | 18

2. Secondary Outcome: Number of Participants With Near-complete Response Rate (≤ 10% Residual Cancer in Primary Tumor Viable)
Time Frame: Post surgery
Population: All participants who have met the eligibility criteria that have signed a consent form and began treatment.
Measure: Number; unit: participants
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Number analyzed (Participants) | 54
participants | 11

3. Secondary Outcome: Percentage of Participants With 3-year Overall Survival
Description: Survival time was defined to be the length of time from start of study therapy to death due to any cause or until last follow-up (censored value).
Time Frame: 3 years
Population: All registered participants who have met the eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Number analyzed (Participants) | 65
percentage of participants | 38.6

4. Secondary Outcome: Percentage of Participants With 2-year Disease-free Survival
Description: Disease-free survival was defined as the time from start of study therapy to documentation of disease recurrence. Participants who died without documentation of recurrence were considered to have had tumor recurrence at the time of death unless there was documented evidence that no recurrence occured before death. Participants who failed to return for evaluation after beginning therapy were censored for recurrence on the last day of therapy. Participants who experienced major treatment violations were censored for recurrence on the date the treatment violation occured.
Time Frame: 2 years
Population: All registered participants who have met the eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Number analyzed (Participants) | 65
percentage of participants | 41.4

5. Secondary Outcome: Number of Participants With Frequent (>=15% Grade 3/4 Incidence) Adverse Events Regardless of Attribution
Description: Adverse events were assessed by NCI CTCAE (Common Terminology Criteria for Adverse Events) v3.0. Grade 1= mild, grade 2= moderate, grade 3= severe, grade 4= life-threatening; and grade 5= death.
Time Frame: Week 1, 3, 5, 7, 9, 4-6 weeks after therapy and within 30 days post surgery
Population: All recruited participants.
Measure: Number; unit: participants
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Number analyzed (Participants) | 70
participants
  Hemoglobin | 12
  Lymphocytes | 30
  Neutrophils | 12
  Dehydration | 13
  Esophagitis | 13
  Nausea | 11

ADVERSE EVENTS:
Arm/Group | Docetaxel + Cisplatin + Panitumumab + RT
Serious Adverse Events (participants affected / at risk) | 46/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + Cisplatin + Panitumumab + RT (N=70)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (12)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Anal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Esophageal fistula (Gastrointestinal disorders) | 2 (2)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 7 (8)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
General symptom (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 5 (5)
Pleural infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 3 (3)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative gastrointestinal injury - Esophagus (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bilirubin increased (Investigations) | 2 (2)
Cardiac troponin I increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (3)
Leukocyte count decreased (Investigations) | 8 (9)
Lymphocyte count decreased (Investigations) | 15 (18)
Neutrophil count decreased (Investigations) | 6 (7)
Platelet count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 10 (10)
Serum albumin decreased (Metabolism and nutrition disorders) | 9 (10)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (5)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (5)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Thrombosis (Vascular disorders) | 10 (13)
Visceral arterial ischemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + Cisplatin + Panitumumab + RT (N=70)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 39 (139)
Hemolysis (Blood and lymphatic system disorders) | 4 (4)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (8)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Cardiac disorder (Cardiac disorders) | 2 (2)
Conduction disorder (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 3 (12)
Diplopia (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (2)
Eyelid function disorder (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Watering eyes (Eye disorders) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (14)
Anal exam abnormal (Gastrointestinal disorders) | 2 (5)
Ascites (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (32)
Diarrhea (Gastrointestinal disorders) | 37 (76)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 12 (27)
Dysphagia (Gastrointestinal disorders) | 30 (49)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 13 (22)
Esophageal pain (Gastrointestinal disorders) | 4 (7)
Esophagitis (Gastrointestinal disorders) | 36 (77)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (18)
Gingival pain (Gastrointestinal disorders) | 2 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 8 (11)
Nausea (Gastrointestinal disorders) | 49 (125)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 28 (44)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 7 (10)
Edema limbs (General disorders) | 4 (6)
Fatigue (General disorders) | 50 (162)
Fever (General disorders) | 7 (10)
General symptom (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 11 (22)
Cytokine release syndrome (Immune system disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 13 (16)
Bronchitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 5 (7)
Opportunistic infection (Infections and infestations) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 9 (14)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 17 (24)
Alkaline phosphatase increased (Investigations) | 10 (20)
Aspartate aminotransferase increased (Investigations) | 19 (25)
Bilirubin increased (Investigations) | 8 (12)
Creatinine increased (Investigations) | 15 (21)
INR increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 3 (22)
Leukocyte count decreased (Investigations) | 56 (156)
Lymphocyte count decreased (Investigations) | 29 (79)
Neutrophil count decreased (Investigations) | 18 (30)
Platelet count decreased (Investigations) | 40 (91)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 19 (30)
Anorexia (Metabolism and nutrition disorders) | 30 (67)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 30 (73)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 20 (29)
Serum albumin decreased (Metabolism and nutrition disorders) | 28 (85)
Serum calcium decreased (Metabolism and nutrition disorders) | 23 (49)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 36 (90)
Serum magnesium increased (Metabolism and nutrition disorders) | 8 (9)
Serum phosphate decreased (Metabolism and nutrition disorders) | 9 (17)
Serum potassium decreased (Metabolism and nutrition disorders) | 18 (31)
Serum potassium increased (Metabolism and nutrition disorders) | 10 (12)
Serum sodium decreased (Metabolism and nutrition disorders) | 16 (35)
Serum sodium increased (Metabolism and nutrition disorders) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (11)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (22)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 16 (28)
Headache (Nervous system disorders) | 3 (4)
Neurological disorder NOS (Nervous system disorders) | 3 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 22 (56)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 13 (36)
Tremor (Nervous system disorders) | 2 (3)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 10 (37)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (8)
Insomnia (Psychiatric disorders) | 11 (38)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 4 (4)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (41)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (30)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (14)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (22)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 33 (82)
Rash acneiform (Skin and subcutaneous tissue disorders) | 66 (279)
Rash desquamating (Skin and subcutaneous tissue disorders) | 26 (60)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 11 (15)
Phlebitis (Vascular disorders) | 2 (3)
Thrombosis (Vascular disorders) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes